CLINICAL TRIAL: NCT01180972
Title: Effects of Environmental Opportunities and Barriers on Physical Activity, Fitness, and Health in Hispanic Children in Wisconsin
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: M-2010-1159
Record Dates: First submitted 2010-08-11; First posted 2010-08-13 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2012-10

CONDITIONS: Obesity, Diabetes, Nutrition, Physical Health
Keywords: Obesity, diabetes, hispanic, physical activity, nutrition
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a pilot community-based research study to examine the effects of specific environmental and social factors on physical activity, fitness, and health of middle school Hispanic children living in an inner-city community.

DETAILED DESCRIPTION:
Our primary hypothesis is that the disparity between a community's potential for physical activity and nutrition, and the realized fitness and health of its children, can be attributed to specific environmental and social factors. "Built environment" studies to date have measured potential for physical activity but have not looked at how social factors mediate an individual's activity within a particular environment. The unique aspect of this proposal is the development of a model that explains how physical, social, cultural, and nutritional SEM layers interact to create gaps between potential and realized physical activity. This project will utilize novel technologies to:

1. identify and analyze characteristics of the social and built environment that inhibit or enhance physical activity and healthy nutrition;
2. determine the direction and extent of influence of these variables on children's activity, nutrition, and health;
3. gather ideas from students, parents, and school staff to inform a potential health campaign to reduce and prevent obesity in the community.

To address these goals and demonstrate a causal relationship between physical activity and the social-nutritional factors within a built environment, the following specific objectives/aims are being addressed:

Specific Aim 1: Assess the built environment for energy requirements of movement, nutrition options, suitability for outdoor physical activity, and for children's actual physical activity and energy expenditure within those environments.

Specific Aim 2: Assess the impact of children's social environment on movement and nutrition choices within the built environment.

Specific Aim 3: Conduct a quantitative assessment of children's fitness, obesity, and indicators of metabolic health.

Specific Aim 4: Develop a quantitative model from Specific Aims 1-3 that describes the causal relationships among children's physical health, community "healthfulness," and other mediating factors such as attitudes, perceptions, and behavior.

ELIGIBILITY:
Inclusion Criteria:

1. The child is in academic attendance at the BGCS in Grades 5-8 and Cherokee Middle School in Grades 6-8.
2. The child and parent or legal guardian is able to provide assent and/or consent.
3. The child is able to understand instructions for study-related activities and comply

Exclusion Criteria:

1. The child is not in academic attendance at the BGCS in Grades 5-8 or at Cherokeed Middle School grades 6-8
2. The child and parent or legal guardian is not able to provide assent and/or consent.
3. The child is able to not able to understand instructions for study-related activities and comply

   -

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Middle - school age children in grades 5-8
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2010-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Assess the built environment for energy requirements of movement, nutrition options, suitability for outdoor physical activity, and for children's actual physical activity and energy expenditure within those environments. | 9/2010 to 3/5/13
  Assess the built environment for energy requirements of movement, nutrition options, suitability for outdoor physical activity, and for children's actual physical activity and energy expenditure within those environments.
  To address this specific aim, we attempt to answer these 2 questions through direct participation from the students and then indirectly through a geographic analysis of the area of interest:
  1. How does the built environment influence children's physical activity, access to healthy food, and individual health and fitness?
  2. Do these relationships vary spatially (e.g., across and within neighborhoods)?

SECONDARY OUTCOMES:
Assess the impact of children's social environment on movement and nutrition choices within the built environment. | 9/2013-3/5/2013
  Data collection is a three step process to analyze the built environment to determine its suitability for walking, bicycling, or other non-motorized means between children's homes, schools, and other common neighborhood destinations. This analysis does not involve direct interaction with or data collection from the students or the parents/legal guardian but will use the children's addresses, zip codes, and the data collected via GPS for Part 1 of this aim.

OTHER OUTCOMES:
Conduct a quantitative assessment of children's fitness, obesity, and indicators of metabolic health. | 9/2013 -03-5/2013
  This aim provides a quantitative assessment of adiposity, cardiovascular fitness, and insulin sensitivity (metabolic factors tied to diabetes risk). These data will be correlated with the physical and nutritional environment.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Carrel, MD, Principal Investigator — UW - Madison - Department of Pediatrics
Locations (1):
- United Community Center/Bruce Guadalupe Community School and Cherokee Middle School, Milwaukee and Madison, Wisconsin, United States